CLINICAL TRIAL: NCT04771650
Title: Addressing Alcohol-Use Related Health Disparities: A Hybrid Effectiveness Implementation Study of a Culturally Adapted MI for Latino/a Alcohol and Drug Users
Brief Title: A Hybrid Effectiveness Implementation Study of Latino/a Alcohol and Drug Users
Acronym: CAMI-HI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Brown University (Other); National Institutes of Health (NIH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Christina Lee, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5688; 1R01AA028507 (NIH)
Record Dates: First submitted 2021-02-11; First posted 2021-02-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Drug Use; Psychological Distress
Keywords: Alcohol; Drug; Latinx; Treatment; Psychological distress
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Clinical effectiveness trial that tests two conditions (CAMI plus booster + standard care compared to assessment + standard care). Health outcomes are reduced drinking, related harms and improvement of mental health. Follow-up at 3,6, and 12 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomized to one of two conditions. They will be unaware of their randomization condition. The Research assistant conducting follow-ups will be unaware of the participant's treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAMI/CAMI booster (Experimental): Culturally Adapted Motivational Interview. Participants will receive a single session, 75 minute addiction counseling discussion that focuses on the causes of addictive behavior. They will receive a CAMI booster session at 2 months and standard care in a primary care setting.
  Interventions: Other: CAMI
- Control (No Intervention): Assessment plus standard care. Participants will complete an assessment, including measures on drinking and drug use. They will also receive standard care in a primary care setting.

INTERVENTIONS:
Other: CAMI — The CAMI is a culturally adapted motivational interview. It is a single 75 minute session that focuses on promoting motivation to change drinking and drug use behavior.
  Arms: CAMI/CAMI booster

SUMMARY:
Alcohol use is a significant problem among Latinxs and immigration-related stress increases risk for substance use. A theoretically-based cultural adaptation of motivational interviewing (CAMI) that specifically integrated discussion of immigration-related stressors (e.g., stigma, social isolation) resulted in significant reductions in alcohol-related harms for those Latinx heavy drinkers with high discrimination compared to standard MI, and reduced anxiety and depressive symptoms one year later compared to MI. Rigorous tests that examine theoretically-informed adaptation of efficacious addiction interventions are not common, yet are needed to advance implementation science. This Hybrid Type 1 Effectiveness-Implementation study will investigate the feasibility of implementing CAMI in a real-world clinical setting. The key questions are: Would CAMI have positive effects among individuals who use both drugs and alcohol? How do providers view this intervention? The investigators will collaborate with a primary care center that serves a mainly Latinx client population to train their Community Wellness Advocates (CWAs) to deliver CAMI to patients who are heavy drinkers. The investigators will conduct a concurrent investigation on the process of implementing CAMI in primary care - a two-arm randomized clinical effectiveness trial will enroll Latinx heavy drinkers (18 years or older) in primary care who use alcohol (and may use other drugs) - and follow them for 12 months after the intervention. Specific Aims are: (1) To examine the impact of CAMI plus a booster session (vs. assessment only) on outcomes: % heavy drinking days, frequency of alcohol-related consequences, depressive/anxiety symptoms, and number of illicit drug use days, using a Hybrid Type 1 Effectiveness-Implementation design and (2) To gather indicators of implementation outcome from multiple stakeholders using a mixed-methods approach. The investigators will follow Curran's framework to evaluate the process of implementation and Proctor's framework to measure implementation outcomes. This study, a first to examine the acceptability of culturally-adapted addiction treatments in primary care settings, will answer essential questions on implementing evidence-based care for Latinxs that can improve health disparities related to substance use. Long term goals are to translate the lessons from this Hybrid study to the broader community to focus on population health for all primary care patients.

DETAILED DESCRIPTION:
Alcohol use is a significant problem among Latinxs because of the disproportionate burden of physical harms and negative consequences associated with substance use relative to other racial/ethnic groups. Factors associated with the stress related to being an immigrant increase risk for substance use. A theoretically-based cultural adaptation of motivational interviewing (CAMI) that specifically integrated discussion of stressors related to immigration (e.g., discrimination, stigma, social isolation) resulted in significant reductions in harms related to alcohol for those Latinx heavy drinkers with high discrimination compared to standard MI, and reduced anxiety and depressive symptoms one year later compared to MI. Rigorous tests that examine theoretically-informed adaptation of efficacious interventions for addictions are not common, yet are needed to advance implementation science because they address questions that are the basis for successful implementation. The proposed Hybrid Type 1 Effectiveness-Implementation study is an important next step in this line of research, which is to investigate the feasibility of implementing the CAMI intervention in a real-world clinical setting. The key questions are: Would CAMI have positive effects among individuals who use both drugs and alcohol? How do providers view this intervention? The investigators will collaborate with a primary care center that serves a mainly Latinx client population to train their Community Wellness Advocates (CWAs) to deliver the CAMI to patients who are heavy drinkers. The investigators will conduct a concurrent investigation on the process of implementing the CAMI in primary care - a two-arm randomized clinical effectiveness trial will enroll Latinx heavy drinkers (18 years or older) in primary care who use alcohol (and may use other drugs) - and follow them for 12 months after the intervention. Specific Aims are: (1) To examine the impact of CAMI plus an in- person booster session (vs. assessment only) on outcomes: % heavy drinking days, frequency of alcohol- related consequences, depressive/anxiety symptoms, and number of illicit drug use days, using a Hybrid Type 1 Effectiveness-Implementation design and (2) To gather indicators of implementation outcome from multiple stakeholders using a mixed-methods approach. The investigators will follow Curran's framework to evaluate the process of implementation and Proctor's framework to measure implementation outcomes: acceptability, adoption, intervention appropriateness, feasibility, overall cost (i.e., CAMI vs. assessment only), and treatment fidelity. This study, a first to examine the acceptability of culturally-adapted addiction treatments in primary care settings, will answer essential questions on implementing evidence-based care for Latinxs that can improve health disparities related to substance use. Long term goals are to translate the lessons from the proposed Hybrid study to the broader community to focus on population health for all primary care patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for binge drinking in the past month (> 4/5 (females/males) drinks/occasion, 1+ days/month)
* Age 18 or older
* Identify as Latinx
* First or second-generation immigrant

Exclusion Criteria:

* Current psychotic symptoms
* Cognitive impairment
* Currently in psychosocial treatment for alcohol use disorder
* Patients who have been enrolled in the Complex Care Management (CCM) before January 1, 2021.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent heavy drinking days | 3 month follow-up
  % heavy drinking days (4 or 5 drinks/day female/male, respectively)
Alcohol-related consequences | 3 month follow-up
  Frequency of alcohol related consequences (e.g., driving under the influence).
Percent drug use days | 3 month follow-up
  % drug use days

SECONDARY OUTCOMES:
Percent heavy drinking days | 6 month follow-up
  % heavy drinking days (4 or 5 drinks/day female/male, respectively)
Percent heavy drinking days | 12 month follow-up
  % heavy drinking days (4 or 5 drinks/day female/male, respectively)
Alcohol-related consequences | 6 month follow-up
  Frequency of alcohol related consequences (e.g., driving under the influence).
Alcohol-related consequences | 12 month follow-up
  Frequency of alcohol related consequences (e.g., driving under the influence).
Center for Epidemiological Studies - Depression | 3 month follow-up
  Level of depressive symptomatology in the past week.
Center for Epidemiological Studies - Depression | 6 month follow-up
  Level of depressive symptomatology in the past week.
Center for Epidemiological Studies - Depression | 12 month follow-up
  Level of depressive symptomatology in the past week.
Beck Anxiety Inventory | 3 month follow-up
  Level of anxiety symptomatology in the past week.
Beck Anxiety Inventory | 6 month follow-up
  Level of anxiety symptomatology in the past week.
Beck Anxiety Inventory | 12 month follow-up
  Level of anxiety symptomatology in the past week.
Percent drug use days | 6 month follow-up
  % drug use days
Percent drug use days | 12 month follow-up
  % drug use days

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Lee, PhD, Principal Investigator — Boston University
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CS, Colby SM, Magill M, Almeida J, Tavares T, Rohsenow DJ. A randomized controlled trial of culturally adapted motivational interviewing for Hispanic heavy drinkers: Theory of adaptation and study protocol. Contemp Clin Trials. 2016 Sep;50:193-200. doi: 10.1016/j.cct.2016.08.013. Epub 2016 Aug 24. PMID 27565832
- [Background] Lee CS, Colby SM, Rohsenow DJ, Martin R, Rosales R, McCallum TT, Falcon L, Almeida J, Cortes DE. A randomized controlled trial of motivational interviewing tailored for heavy drinking latinxs. J Consult Clin Psychol. 2019 Sep;87(9):815-830. doi: 10.1037/ccp0000428. PMID 31403817